CLINICAL TRIAL: NCT01274208
Title: Enhanced HCV Nonstructural Protein 3 (NS3) -Specific T Cell Proliferation,Interferon γ (IFNγ) and Interleukin-10 (IL-10) Secreting Clones, and Peripheral Blood Natural Killers T Cells ( NKT Cells) in Patients With Type I Gaucher Disease Infected With HCV : An Advantage in Anti Hepatitis Immunity?
Brief Title: Examining the Immune Response in Patients With Gaucher Disease and Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Ari Zimran, Prof. Ari Zimran, Shaare Zedek Medical Center
Other Study IDs: SZMC- 89/10
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Gaucher Disease; Hepatitis C
Keywords: Gaucher disease, Hepatitis C , Glucocerebroside immunity
MeSH Terms: conditions — Gaucher Disease; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gaucher Disease with Hepatitis C

SUMMARY:
Study objectives:

* Investigate the anti-HCV response in patients with Gaucher disease(GD)
* Define the potential role of high levels of Glucocerebroside in the immune system

Study hypothesis:

High levels of Glucocerebroside can be used as a tool in the antiviral treatment of hepatitis C by potentiating the immune response of natural killer T cells and dendritic cells

DETAILED DESCRIPTION:
Gaucher disease is the most common glycolipid storage disorder, caused by reduced activity of the lysosomal enzyme glucocerebrosidase, which leads to the accumulation of the substrate, glucocerebroside (GC), in the cells of the reticulo-endothelial system.

One of the hallmarks of GD is its great phenotypic heterogeneity with variable presentations and symptoms, beginning with a lethal variant of infants dying at or near birth with hydrops fetalis and ichthyoids at one extreme and totally asymptomatic individuals without any physical or laboratory abnormalities at the other extreme.

This autosomal recessive disease is pan-ethnic, but it is especially prevalent among Ashkenazi Jews. From over 300 different mutations reported in the glucocerebrosidase gene, five account for 98% of the disease-producing alleles. Of these mutations, N370S (or 1226G) occurs in 1 out of 17 Ashkenazi individuals, leading to a disease frequency of 1:850 in this ethnic group.

The high prevalence of more than a single mutation among Ashkenazi Jews and the existence of two additional rare inherited lysosomal glycolipid storage diseases, Tay Sachs and Nieman Pick, at a higher prevalence within the same ethnic group is believed to be caused by selective advantage.

Available genetic data are consistent with a founder effect(4) whereas the nature of such an advantage has not been identified.

The aim of this study was to investigate the anti-HCV immune response in patients with GD in an attempt to define the potential role of high levels of GC in the immune system and antiviral immunity.

Study importance:

The host metabolic background exerts a profound effect on antiviral immunity, which may influence the clinical course of chronic HCV infection.

The accumulation of GC in patients with GD may provide a selective evolutionary advantage to these patients.

Glucocerebroside was recently tested in human trials and shown to be effective in altering NKT- dependent metabolic pathways, insulin resistance, and associated liver injury.

The present study examine the capability of Glucocerebroside to be be used as a tool in the antiviral treatment of hepatitis C by potentiating the immune response of natural killer T cells and dendritic cells.

Statistical Analysis:

Data are presented as the mean ± standard deviation (SD). The Kruskal Wallis non-parametric ANOVA test was used to identify differences between the study groups.

The student t-test and non-parametric Mann-Whitney test were used to compare quantitative variables between the study groups as appropriate; P <0.05 was considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Gaucher disease
* Patients with hepatitis C without Gaucher disease
* Individuals or patients without Gaucher disease and hepatitis C
* Individuals or patients who signed an approval for the research
* Men and women 18< years of age , pregnant women

Exclusion Criteria:

* Inabillity to give an approval for the research
* Acute liver disease that can alter the lab results , such as: Rt. congestive heart failure

severe infection ,inflammation, medication such as : Statins , Isoniazid ,

Amiodarone

- Patients who received treatment for hepatitis C such as: Interferon ,

Pegylated interferon , Ribavirin

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Gaucher Disease were recruited from the Sha'are Zedek Gaucher disease clinic, a national referral center for the disease.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Gaucher patients' immune system provide enhanced immunity against hepatitis c virus | 6 months

SECONDARY OUTCOMES:
the role Glucocerebroside level have by enhanced immunity in patients with Gaucher disease | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Melamud, Dr., Principal Investigator — Gaucher Clinic , Shaare zedek Hospital
Locations (2):
- Israel (2):
  - Shaare Zedek , Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem

REFERENCES:
- [Background] Elstein D, Abrahamov A, Hadas-Halpern I, Zimran A. Gaucher's disease. Lancet. 2001 Jul 28;358(9278):324-7. doi: 10.1016/S0140-6736(01)05490-3. No abstract available. PMID 11498237
- [Background] Butters TD. Gaucher disease. Curr Opin Chem Biol. 2007 Aug;11(4):412-8. doi: 10.1016/j.cbpa.2007.05.035. Epub 2007 Jul 23. PMID 17644022
- [Background] Beutler E. Gaucher disease: multiple lessons from a single gene disorder. Acta Paediatr Suppl. 2006 Apr;95(451):103-9. doi: 10.1111/j.1651-2227.2006.tb02398.x. PMID 16720474
- [Background] Slatkin M. A population-genetic test of founder effects and implications for Ashkenazi Jewish diseases. Am J Hum Genet. 2004 Aug;75(2):282-93. doi: 10.1086/423146. Epub 2004 Jun 18. PMID 15208782
- [Background] Beutler E. Gaucher disease as a paradigm of current issues regarding single gene mutations of humans. Proc Natl Acad Sci U S A. 1993 Jun 15;90(12):5384-90. doi: 10.1073/pnas.90.12.5384. PMID 8516282
- [Result] Zigmond E LG, Pappo O, Zangen S, Levy Sklair M, Hemed N, Rabbani E, Itamar R, Ilan Y, Margalit M. Treatment of non-alcoholic steatohepatitis by B-glucosylceramide: A phase I/II clinical study. Hepatology 2006;44 .180A, .